CLINICAL TRIAL: NCT06964373
Title: Cervical Ripening Balloon for Same-Day Cervical Preparation for Second Trimester Termination
Brief Title: Cervical Ripening Balloons for Same-Day Cervical Prep
Acronym: CRB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-493
Record Dates: First submitted 2025-04-07; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Dilation and Evacuation
MeSH Terms: conditions — Dilatation, Pathologic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cervical Ripening Balloon (Experimental)
  Interventions: Device: Cervical Ripening Balloon
- Osmotic Dilators (Active Comparator)
  Interventions: Device: Osmotic Dilators

INTERVENTIONS:
Device: Cervical Ripening Balloon — 30 milliliter Foley balloon
  Arms: Cervical Ripening Balloon
Device: Osmotic Dilators — Dilapan-S
  Arms: Osmotic Dilators

SUMMARY:
The goal of this clinical trial is to learn if a cervical ripening balloon (Foley balloon) works to prepare the cervix before same-day outpatient dilation and evacuation (D&E). The main questions it aims to answer are:

* Is cervical preparation with cervical ripening balloon for same-day outpatient D&E non-inferior to cervical preparation with osmotic dilators?
* How feasible and safe is cervical preparation with cervical ripening balloon for same-day outpatient D&E?
* How acceptable is cervical preparation with cervical ripening balloon for same-day outpatient D&E?

Participants will:

* Have cervical preparation with cervical ripening balloon (experimental group) or osmotic dilators (usual care group)
* Complete two surveys, one about the cervical preparation and one about the D&E procedure

ELIGIBILITY:
Inclusion Criteria:

* Individuals who desire outpatient dilation and evacuation (D&E)
* At least 18 years of age
* Able and willing to consent
* Gestational duration between 18 weeks 0 days and 19 weeks 6 days as determined by ultrasound
* Able to read and understand English or Spanish
* Able to obtain reliable post-procedure transportation
* Able to observe fasting guidelines of 6 hours prior to the D&E procedure

Exclusion Criteria:

* Medical conditions that require procedural management in the operating room
* Preference for D&E procedure in the operating room

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
D&E procedure length (minutes) | during procedure
  From insertion of first instrument to removal of speculum

SECONDARY OUTCOMES:
Starting dilation (French gauge) | during procedure
  Pratt dilator size in French gauge (sequential numbered instruments with size corresponding to diameter)
Additional dilation (French gauge) | during procedure
  Pratt dilator size in French gauge (sequential numbered instruments with size corresponding to diameter)
Estimated blood loss (milliliters) | during procedure
  Amount of blood loss, measured in milliliters throughout the procedure
Additional sedation medication administered | during procedure
  yes/no
Pain (Visual Analog Scale) | during procedure
  10 point visual analog scale with values from 0-10, with 0 being "No pain" and 10 being "Worst possible pain." Electronic slider measure so participants can specify up to 0.001 value.
Administration of uterotonic medications | during procedure
  yes/no
Cervical laceration | during procedure
  yes/no
Estimated blood loss > 500 milliliters | From enrollment to 24 hours after enrollment
  yes/no
Hospital transfer | From enrollment to 24 hours after enrollment
  yes/no
Feasibility of cervical preparation (physician-reported) | From enrollment to 24 hours after enrollment
  Yes/ No: "Is this type of cervical prep feasible for future patients" and qualitative free-text responses
Likelihood to recommend cervical preparation (participant-reported) | From enrollment to 24 hours after enrollment
  Modified Likert scale: Very unlikely, Somewhat unlikely, Neither likely nor unlikely, Somewhat likely, Very likely
Acceptability of cervical preparation (physician-reported) | From enrollment to 24 hours after enrollment
  Yes/ No: "Is this type of cervical prep acceptable for future patients" and qualitative free-text responses
Satisfaction with level of pain management (participant-reported) | From enrollment to 24 hours after enrollment
  Yes/ No: "Are you satisfied with your level of pain management..." and qualitative free-text responses

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States